CLINICAL TRIAL: NCT02956720
Title: Clinical Evaluation of UltraShape Power System in Conjunction With the U-Sculpt-N Transducer for Non-invasive Circumference Reduction
Brief Title: UltraShape Power in Combination With U-sculpt-n Transducer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Syneron Candela (Industry)
Responsible Party: Principal Investigator, Ronen Glesinger, Principal investigator, Syneron Candela
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF21321
Record Dates: First submitted 2016-10-30; First posted 2016-11-07 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Circumference Reduction

STUDY DESIGN:
Intervention Model Description: prospective, single arm

ARMS (1):
- single arm (Experimental)
  Interventions: Device: UltraShape Power

INTERVENTIONS:
Device: UltraShape Power — non-invasive body contouring procedure

SUMMARY:
Prospective, open label, self - controlled, single arm, clinical study to assess the performance of the UltraShape Power using the U-Sculpt-N on outer thigh and/or flank for circumference reduction versus self-control.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥18 and ≤60 years of age at the time of enrollment
2. Fat thickness of at least 1.5 cm in the outer thigh and/or flank (measured by calibrated caliper)
3. For women of child-bearing potential: negative urine pregnancy test
4. General good health confirmed by medical history and skin examination of the treated area
5. Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed.

Exclusion Criteria:

1. History of un-balanced hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator
2. Current hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease
3. Having a permanent implant in the treated area, such as metal plates, or an injected chemical substance such as silicone
4. Previous liposuction in the treatment areas within 12 months
5. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing
6. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months
7. Childbirth within the last 12 months or women who are breastfeeding a child

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Outer thigh circumference reduction | up to 24 week
  To evaluate circumference reduction of outer thigh post treatment with UltraShape Power device used with the U-Sculpt-N transducer versus control side.
Treatment-related adverse events | up to 24 week
  The frequency and severity of all treatment-related adverse events during and after using the UltraShape Power device used with the U-Sculpt-N transducer.

SECONDARY OUTCOMES:
Subject satisfaction questionnaire | up to 24 week
  The assessment of subject satisfaction with treatment will be recorded during relevant visits (starting following the first treatment) using a 5-point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Beit Noah, Ramat Gan, Israel